CLINICAL TRIAL: NCT03035929
Title: Diagnosing Natriuretic Peptide Deficiency: A Pilot Study
Brief Title: Diagnosing Natriuretic Peptide Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Katherine N. Bachmann, MD, Instructor in Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 161482
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Healthy; Lean
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy (Experimental): 10 Healthy subjects will undergo study procedures at four study visits.
  All subjects will undergo the same procedures and interventions.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — A single dose of dexamethasone IV 4 mg will be administered.
  Other Names: Dexamethasone IV

SUMMARY:
In this pilot study, the investigators will determine the response of the natriuretic peptide (NP) hormone system after a dose of intravenous dexamethasone (a steroid medication). The goal of the proposed project is to generate preliminary data that will be used to develop power calculations, inform cutoff ranges, and inform the timing of the NP response for larger subsequent studies.

Aim: To determine the range of distribution and time course of natriuretic peptide (NP) responses to a single dose of dexamethasone IV 4 mg in healthy lean individuals.

Hypothesis: Determination of the NP responses (the range and time course of changes in NP levels) to dexamethasone in 10 healthy individuals will inform the time course and frequency of blood sampling in a definitive prospective study, as well as enable investigators to perform a sample size calculation for a definitive prospective study.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion criteria:

* Men and women ages 18-50 years
* BMI 18.5 to <25 kg/m^2

Exclusion Criteria:

* Significant use of systemically-absorbed glucocorticoids currently or for an extended period of time during the prior 6 months
* Current use of antihypertensive medications
* Current use of metformin, or any antidiabetic medications (which could affect glucose and insulin levels)
* Current use of medications known to affect dexamethasone metabolism, including phenytoin, rifampin, carbamazepine, troglitazone, and barbiturates
* Active, clinically significant infection at time of visit
* History of adrenal insufficiency or Cushing's syndrome
* Prior or current cardiovascular disease, renal disease, or liver disease
* Diabetes mellitus, pre-diabetes, impaired fasting glucose, or impaired glucose tolerance
* Atrial fibrillation
* Bleeding disorder or anemia
* Elevated Liver Functions Tests > 2 times upper limit of normal
* Estimated glomerular filtration rate < 60 ml/min
* HbA1c > 5.7
* Abnormal sodium or potassium level
* Positive pregnancy test, women of child-bearing age not practicing birth control, women who are breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine N Bachmann, MD, Principal Investigator — Vanderbilt Endocrinology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant withdrew after consent but before the baseline visit and is not included in the results.
Groups:
- Healthy: Healthy subjects will be enrolled and each will undergo study procedures at four study visits.
  All subjects will undergo the same procedures and interventions.
  Dexamethasone: A single dose of dexamethasone IV 4 mg will be administered.
Period: Overall Study
Arm/Group | Healthy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy: Healthy subjects will be enrolled and each will undergo study procedures at 4 study visits.
  All subjects will undergo the same procedures and interventions.
  Dexamethasone: A single dose of dexamethasone IV 4 mg will be administered.
Arm/Group | Healthy
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27.5 [24.5 to 29.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in NT-proANP From Baseline to 8 Hours
Description: Change in natriuretic peptide levels after drug administration
Time Frame: baseline and 8 hours
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Healthy
Number analyzed (Participants) | 10
nmol/l | -0.33 (0.25)

2. Primary Outcome: Changes in NT-proBNP From Baseline to 8 Hours
Description: Change in natriuretic peptide levels after drug administration
Time Frame: Baseline and 8 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Healthy
Number analyzed (Participants) | 10
pg/ml | 18.4 (20.3)

3. Secondary Outcome: Changes in NT-proANP
Description: Change in natriuretic peptide levels after drug administration from baseline to 24 hours, 48 hours, and 72 hours
Time Frame: baseline, 24 hours, 48 hours and 72 hours
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Healthy
Number analyzed (Participants) | 10
nmol/l
  Change from baseline to 24 hours | -0.23 (.22)
  Change from baseline to 48 hours | 0.17 (.36)
  Change from baseline to 72 hours | -0.05 (.33)

4. Secondary Outcome: Changes in NT-proBNP
Description: Change in natriuretic peptide levels after drug administration from baseline to 24 hours, 48 hours, and 72 hours
Time Frame: at baseline, 24 hours, 48 hours and 72 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Healthy
Number analyzed (Participants) | 10
pg/ml
  Change from baseline to 24 hours | -5.0 (26.9)
  Change from baseline to 48 hours | -23.4 (41.4)
  Change from baseline to 72 hours | -16.9 (39.6)

5. Secondary Outcome: BNP (B-type Natriuretic Peptide)
Description: Natriuretic peptide levels after drug administration
Time Frame: 0-8 hrs, 24 hrs, 48 hrs, 72 hrs after drug administration
Population: Analysis was not able to be completed on any of the samples because reliable assay is not available at this time.
Arm/Group | Healthy
Number analyzed (Participants) | 0

6. Secondary Outcome: ANP (Atrial Natriuretic Peptide)
Description: Natriuretic peptide levels after drug administration
Time Frame: 0-8 hrs, 24 hrs, 48 hrs, 72 hrs after drug administration
Population: Analysis was not able to be completed on any of the samples because reliable assay is not available at this time.
Groups:
- Healthy: 10 Healthy subjects will be enrolled and each will undergo study procedures at 4 study visits.
  All subjects will undergo the same procedures and interventions.
  Dexamethasone: A single dose of dexamethasone IV 4 mg will be administered.
Arm/Group | Healthy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 48 hours
Groups:
- Healthy: Healthy subjects will be enrolled and each will undergo study procedures at three study visits.
  All subjects will undergo the same procedures and interventions.
  Dexamethasone: A single dose of dexamethasone IV 4 mg will be administered.
Arm/Group | Healthy
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy (N=10)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03035929/Prot_SAP_000.pdf